CLINICAL TRIAL: NCT05696834
Title: Sclerotherapy With Adjuvant Bone Marrow Injection In Management of Aneurysmal Bone Cyst
Brief Title: Sclerotherapy and Bone Marrow Injection In Aneurysmal Bone Cyst
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdallah Mousa Elwany Hassan, principal investigator, Al-Azhar University
Other Study IDs: SABMIMABC
Record Dates: First submitted 2023-01-08; First posted 2023-01-25 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Sclerotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sclerotherapy and bone marrow: Sclerotherapy With Adjuvant Bone Marrow Injection In Management of Aneurysmal Bone Cyst
  Interventions: Procedure: Sclerotherapy With Adjuvant Bone Marrow Injection In Management of Aneurysmal Bone Cyst

INTERVENTIONS:
Procedure: Sclerotherapy With Adjuvant Bone Marrow Injection In Management of Aneurysmal Bone Cyst — Sclerotherapy With Adjuvant Bone Marrow Injection In Management of Aneurysmal Bone Cyst

SUMMARY:
Aneurysmal bone cysts (ABCs) are benign, locally destructive growing bone tumors, which were first described in 1942 by Jaffé and Lichtenstein (1). They are most often diagnosed in childhood and early adulthood. The literature reports that ABCs comprise 1-6% of all primary benign bone tumors (2). Most cases of ABCs (75-90%) are reported for patients younger than 20 years, with a slightly higher incidence for females (3). Most common localizations are the pelvis, the metaphysis of long bones and the spine, but ABCs can also affect any other localization(2). ABCs that are associated with a preexisting osseous lesion are defined as secondary ABCs. They represent approximately 30% of all ABCs (2). Secondary ABCs can occur, e.g., in cases of a giant cell tumor, chondroblastoma or telangiectatic osteosarcoma

DETAILED DESCRIPTION:
The clinical symptoms of an ABC are usually accidently discovered or may consist of pain and swelling in the affected region and pathological fractures ( complete and incomplete ) can be observed occasionally. In conventional radiography a relatively well-defined osteolytic, expansile lesion with possible blowout of the periosteum and a soap-bubble appearance can be found (4). MRI scanning shows cystic formations with typical fluid-fluid levels due to blood sedimentation (7). Because of the possible rapid growth with local destruction, the literature describes cases of ABCs that mimic malignant bone tumors

ELIGIBILITY:
Inclusion Criteria:

* All Patients above age of 1 year.
* The affected area was all bones except skull, ribs, and other non-orthopedic specialties.
* Primary or recurrent ABC
* Incomplete Fractured affected bones as greenstick fracture.
* Healed Pathological fracture without any surgical intervention

Exclusion Criteria:

* ABC. In skull, ribs, and other non-orthopedic specialties.
* Age less than 1 year
* Suspected malignancy or other bone cysts
* Complete fractured bones and healed pathological fracture with surgical intervention.

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 20 Patients complaining from pain at all affected bones. All patients undergo to examination and investigated by radiological (Plain X-rays and MRI).
  All patients undergo to C-arm plain X-rays guided biopsy, aspirated histopathology, and Chemical study ( as Alkaline Phosphatase assessment ) as pre-operative planning.
  All patients received an injection of polidocanol intralesional as standard treatment with a dose: 2- 4 mg / Kg .
  Ossification ( healing ) was assessed on plain X-ray, and the pain was evaluated on a visual analog scale (VAS).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Healing | 1 year
  Results will discuss in this study, according to assessment of ABC healing ( complete or not ) , and also following assessment of recurrence rate and incidence of complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Al-Azhar University Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dormans JP, Hanna BG, Johnston DR, Khurana JS. Surgical treatment and recurrence rate of aneurysmal bone cysts in children. Clin Orthop Relat Res. 2004 Apr;(421):205-11. doi: 10.1097/01.blo.0000126336.46604.e1. PMID 15123949
- [Background] Shiels WE 2nd, Mayerson JL. Percutaneous doxycycline treatment of aneurysmal bone cysts with low recurrence rate: a preliminary report. Clin Orthop Relat Res. 2013 Aug;471(8):2675-83. doi: 10.1007/s11999-013-3043-2. Epub 2013 May 14. PMID 23670673